CLINICAL TRIAL: NCT03775629
Title: A Randomized, Open-label, Multiple-dose, Parallel Study to Compare the Pharmacokinetics and to Evaluate Drug-Drug Interaction of "CG100650" in Healthy Volunteers
Brief Title: Drug-Drug Interaction Study of "CG100650" in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CrystalGenomics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CG100650-1-01
Record Dates: First submitted 2018-12-09; First posted 2018-12-14 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Healthy
MeSH Terms: interventions — CG100649; Tramadol

STUDY DESIGN:
Intervention Model Description: Group A: Tramadol hydrochloride +Polmacoxib Group B: Polmacoxib Group C: Tramadol hydrochloride
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Polmacoxib and Tramadol combination (Experimental): Tramadol + Polmacoxib capsule
  Interventions: Drug: Polmacoxib and Tramadol combination
- Polmacoxib (Active Comparator): Polmacoxib
  Interventions: Drug: Polmacoxib
- Tramadol (Active Comparator): Tramadol hydrochloride (HCl)
  Interventions: Drug: Tramadol hydrochloride

INTERVENTIONS:
Drug: Polmacoxib and Tramadol combination — Tramadol hydrochloride , Polmacoxib
  Arms: Polmacoxib and Tramadol combination
Drug: Polmacoxib — Polmacoxib
  Arms: Polmacoxib
Drug: Tramadol hydrochloride — Tramadol hydrochloride (HCl)
  Other Names: Tramadol
  Arms: Tramadol

SUMMARY:
This is a randomized, open-label, multiple-dose, parallel, Phase 1 study to compare the pharmacokinetics and to evaluate Drug-Drug Interaction of "CG100650" in healthy volunteers.

DETAILED DESCRIPTION:
This is a randomized, open label, multiple-dose, parallel study to compare PK and to evaluate Drug-Drug Interaction of CG100650 in healthy volunteers.

Total of 39 health volunteers will be randomized to receive either of Group A, B or C for 14 days (13 subjects each).

[Group A] Tramadol +Polmacoxib capsule [Group B] Polmacoxib capsule [Group C] Tramadol

Pharmacokinetic parameters will be evaluated as primary endpoint by changes from baseline;

Safety evaluation will be carried out by conducting vital sign, laboratory test, ECG, and collecting AE, CM by different Group.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female aged ≥ 19 years and ≤ 50 years
2. Without inborn or chronic disease and no symptoms in physical examination
3. BMI(Body Mass Index) result ≥ 18kg/m 2 and ≤ 30kg/m2
4. Adequate clinical laboratory test results as evidenced by Hematology, Hemostasis, Biochemistry, Urinalysis, Serology and so on
5. Subject who understand the objective, method of the study and the characteristics of investigational drug and expected adverse events and provide written informed consent prior to study participation
6. Negative pregnancy test(hCG) and agree to contraception during the trial

Key Exclusion Criteria:

1. History of hypersensitivity to investigational products
2. History of hypersensitivity or allergic reaction to sulfonamide.
3. Patients with a history of asthma, acute rhinitis, nonspecific polyps, angioedema, urticaria or allergic reactions to aspirin or other nonsteroidal anti- inflammatory analgesics (including COX-2 inhibitors)
4. Genetically galactose intolerance, lactose intolerance or Glucose-Galactose Malabsorption
5. Any other reasons or situations that the investigator decides the patient is not eligible to participate the clinical trial.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
AUCtau of Polmacoxib and Tramadol | up to 4 weeks
Cmax of Polmacoxib and Tramadol | up to 4 weeks

SECONDARY OUTCOMES:
Cmax of Polmacoxib | up to 4 weeks
AUC tau of Polmacoxib | up to 4 weeks
Cmax of Tramadol | up to 4 weeks
AUCtau of Tramadol | up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea